CLINICAL TRIAL: NCT04096235
Title: A Pilot Study to Evaluate the Use of the Neotech RAM Nasal Cannula for CPAP and Bi-PAP Application in Infants 28-42 Weeks Gestation in a Neonatal Intensive Care Unit (NICU)
Brief Title: A Study to Evaluate the Use of the Neotech RAM Nasal Cannula for CPAP and Bi-PAP Application in Infants 28-42 Weeks Gestation in a Neonatal Intensive Care Unit (NICU)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: change in clinical practice
Sponsor: Englewood Hospital and Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E-19-763
Record Dates: First submitted 2019-09-16; First posted 2019-09-19 (Actual); Last update posted 2021-08-20 (Actual); Status verified 2021-08

CONDITIONS: Neonatal Respiratory Distress
MeSH Terms: conditions — Pulmonary Atelectasis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- RAM Cannula (Experimental)
  Interventions: Other: RAM Nasal Cannula

INTERVENTIONS:
Other: RAM Nasal Cannula — The RAM Nasal Cannula is a means of providing CPAP and Bi-PAP to infants 28-42 weeks gestation to prevent nasal septal erosion.

SUMMARY:
This study will explore the RAM Nasal Cannula as a means of providing CPAP and Bi-PAP to infants 28-42 weeks gestation to prevent nasal septal erosion.

ELIGIBILITY:
Inclusion:

* Infants with birth weight < 1500 grams AND/OR <32 weeks gestational age
* Infants between 34-42 weeks gestational age and exclusive breastfeeding with no risk of nasal septal erosion OR Infants between 28-42 weeks gestational age at risk of nasal septal erosion

Exclusion:

* Infants with major congenital and upper airway anomalies
* Infants requiring ETT (endotracheal tube) mechanical ventilation
* Infants receiving no respiratory support

Ages: 28 Weeks to 42 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 14 (Actual)
Dates: Start 2019-10-18 (Actual); Primary Completion 2021-07-08 (Actual); Study Completion 2021-07-08 (Actual)

PRIMARY OUTCOMES:
NCPAP | 5 days
  The study will determine if the RAM Nasal Cannula is providing adequate CPAP to neonates. This will be measured with the Braden Q score. The Braden Q Scale is composed of seven subscales. All seven subscales are rated from 1 (least favorable)to4(most favorable); patients receive only one score per subscale.
Bi-PAP | 5 days
  The study will determine if the RAM Nasal Cannula is providing adequate Bi-PAP to neonates. This will be measured with the Braden Q score every 3 hours. The Braden Q Scale is composed of seven subscales. All seven subscales are rated from 1 (least favorable)to4(most favorable); patients receive only one score per subscale.
NCPAP | 5 days
  The study will determine if the RAM Nasal Cannula is providing adequate CPAP to neonates. This will be measured with SpO2 Level every 3 hours. The SpO2 will be measured in percentage
NCPAP | 5 days
  The study will determine if the RAM Nasal Cannula is providing adequate CPAP to neonates. This will be measured with Pulse Oximetry Level every 3 hours. The pulse oximetry is measured in millimeters
Bi-PAP | 5 days
  The study will determine if the RAM Nasal Cannula is providing adequate Bi-PAP to neonates. This will be measured with SpO2 Level every 3 hours. The SpO2 will be measured in percentage
Bi-PAP | 5 days
  The study will determine if the RAM Nasal Cannula is providing adequate Bi-PAP to neonates. This will be measured with Pulse Oximetry Level every 3 hours. The pulse oximetry is measured in millimeters

SECONDARY OUTCOMES:
High Flow Humidity | 5 days
  The study will determine if the RAM Nasal Cannula administers high flow humidity (>8Ipm) . This will be measured with the Braden Q score, every 3 hours.The Braden Q Scale is composed of seven subscales. All seven subscales are rated from 1 (least favorable)to4(most favorable); patients receive only one score per subscale.
High Flow Humidity | 5 days
  The study will determine if the RAM Nasal Cannula administers high flow humidity (>8Ipm) . This will be measured with Pulse Oximetry Level every 3 hours. The pulse oximetry is measured in millimeters.
High Flow Humidity | 5 days
  The study will determine if the RAM Nasal Cannula administers high flow humidity (>8Ipm) . This will be measured with SpO2 Level every 3 hours. The SpO2 will be measured in percentage

CONTACTS AND LOCATIONS:
Locations (1):
- Englewood Hospital and Medical Center, Englewood, New Jersey, United States